CLINICAL TRIAL: NCT00415948
Title: Myeloperoxidase and Multi-Markers In the Diagnosis of Diagnoses of Acute Coronary Syndrome (MIDAS) - Sample Procurement
Status: Completed | Type: Observational
Sponsor: Abbott RDx Cardiometabolic (Other)
Other Study IDs: BSTE-0101
Record Dates: First submitted 2006-12-21; First posted 2006-12-25 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-12

CONDITIONS: Acute Coronary Syndrome (ACS)
Keywords: Heart; Cardiac; Acute Coronary Syndrome; Sample Procurement
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma Specimens

INTERVENTIONS:
Device: Biomarkers

SUMMARY:
The purpose of the study is to procure blood samples from patients who present to the Emergency Department with suspected ACS (Acute Coronary Syndrome).

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational, and sample procurement study of adult subjects presenting to an Emergency Department (ED) in whom ACS is in the differential diagnosis. Subjects must present to one of the participating EDs within 6 hours or less from the time of symptom onset, and must have experienced at least 30 minutes of chest discomfort. Those ED patients with possible ACS who meet the inclusion/exclusion criteria will be approached for study enrollment by trained research personnel.

The patient's diagnostic work-up and treatment will continue per the standards of the treating institution. As indicated by their clinical presentation, all subjects in the study will have objective cardiac testing for evidence of coronary artery disease (CAD) during or in close proximity to the index ED visit or hospital admission. For this study, objective cardiac testing will consist of one of the following tests: exercise treadmill, coronary angiography, myocardial stress imaging, stress magnetic resonance imaging (MRI), sestamibi scan, or dobutamine echocardiogram. Cardiac events and procedures, such as angioplasty-stenting and coronary artery bypass surgery (CABG), will be recorded during the index ED visit, hospitalization and post-hospital follow-up period. Subjects will have a 30-day and 6-month follow-up contact by phone to collect this information on cardiac events, procedures, and survival.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at time of enrollment
* Patient presenting to the ED within 6 hours or less from symptom (chest discomfort consistent with possible ACS) onset
* Patient experiencing at least 30 minutes of chest discomfort, consistent with possible ACS, from time of symptom onset; patients who have symptoms of shorter duration due to pharmacologic intervention may be included
* Physician plans to perform objective cardiac testing as defined by the protocol

Exclusion Criteria:

* Patient (or legal representative) unable or unwilling to provide informed consent
* Patient (or legal representative) refusal of medical record review or telephone follow-up at 30 days or 6 months
* Patient (or legal representative) refusal of multiple blood sample collection over the study period
* Prisoners or other institutionalized individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting the to the ED within 6 hours with symptoms consistent with ACS.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-12; Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Peacock, MD, Principal Investigator — The Cleveland Clinic
Locations (18):
- United States (18):
  - UC Davis, Sacramento, California
  - Yale University, New Haven, Connecticut
  - St Agnes Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Ingham Regional Medical Center, Lansing, Michigan
  - New York Methodist Hosptial, Brooklyn, New York
  - SUNY Stony Brook, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Virginia, Charlottesville, Virginia
  - Sentara Norfolk General Hopsital, Norfolk, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia